CLINICAL TRIAL: NCT04033432
Title: A Phase II Study of sEphB4-HSA in Metastatic Castration-Resistant Prostate Cancer
Brief Title: sEphB4-HSA in Treating Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: Vasgene Therapeutics, Inc (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 18U10; NCI-2019-03773 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00209511; NU 18U10 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Castration-Resistant Prostate Carcinoma Refractory to Second-Generation Androgen Receptor Axis-Targeted Agents; Metastatic Prostate Adenocarcinoma; Progressive Disease; Prostate Carcinoma Metastatic in the Bone; Prostate Carcinoma Metastatic in the Soft Tissue; PSA Progression; Stage IVB Prostate Cancer AJCC v8; Testosterone Less Than 50 ng/dL
MeSH Terms: conditions — Disease Progression; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (recombinant EphB4-HSA fusion protein) (Experimental): Patients receive recombinant EphB4-HSA fusion protein IV over 60 minutes on day 1. Treatment repeats every 14 days for cycles 1-6 and then every 21 days for subsequent cycles. Patients may continue to receive sEphB4-HSA treatment until no longer clinically benefiting (PCWG3), unacceptable toxicity, treatment delay >= 4 weeks, or prohibitive illness/change in patient?s condition, or patient decides to withdraw from study.
  Interventions: Biological: Recombinant EphB4-HSA Fusion Protein

INTERVENTIONS:
Biological: Recombinant EphB4-HSA Fusion Protein — Given IV
  Other Names: sEphB4-HSA

SUMMARY:
The purpose of this phase II, single-arm, open-label, three center study is to evaluate the efficacy, safety, and tolerability of sEphB4-HSA in patients with mCRPC (metastatic castration-resistant prostate cancer). The study drug, sEphB4-HAS, is a form of protein that has not been approved for sale by the United States Food and Drug Administration (FDA). The study drug prevents tumor cells from multiplying and blocks several compounds that promote the growth of blood vessels that bring nutrients to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the efficacy of recombinant EphB4-HSA fusion protein (sEphB4-HSA) in patients with metastatic castration resistant prostate cancer (mCRPC) as measured by confirmed prostate specific antigen (PSA) response rate.

SECONDARY OBJECTIVES:

I. The safety and tolerability of sEphB4-HSA in patients with mCRPC according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

II. To assess the time to PSA progression. III. To assess overall response rate in patients with measurable disease using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (soft tissue) and Prostate Cancer Working Group 3 (PCWG3) (bone) criteria.

IV. To assess radiological progression free survival (rPFS) using RECIST 1.1 (soft tissue) and PCWG3 (bone) criteria.

EXPLORATORY OBJECTIVES:

I. To explore molecular changes associated with EphB4 and ephrinB2 expression in tumor specimens (primary and/or metastatic tissue).

II. To explore association of response with molecular biomarkers including aberrations in the PI3K pathway, MYC and TP53.

III. To assess immune cell infiltration of tumors in biopsies. IV. To assess circulating immune changes associated with treatment.

OUTLINE:

Patients receive recombinant EphB4-HSA fusion protein intravenously (IV) over 60 minutes on day 1. Treatment repeats every 14 days for cycles 1-6 and then every 21 days for subsequent cycles. Patients may continue to receive sEphB4-HSA treatment until no longer clinically benefiting (PCWG3), unacceptable toxicity, treatment delay >= 4 weeks, or prohibitive illness/change in patient?s condition, or patient decides to withdraw from study.

After completion of study treatment, patients are followed up at 30 days and then every 6 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathologically confirmed diagnosis of prostate adenocarcinoma
* Patients must have metastatic (M1) disease as evidenced by soft tissue and/or bony metastases on computed tomography (CT) or magnetic resonance imaging (MRI) scan or technetium bone scan
* Patients must have castration resistant disease with disease progression despite castrate levels of testosterone (testosterone =< 50 ng/dL)
* Patients must have received and progressed on at least one second generation androgen receptor (AR) targeted therapy for castration resistant disease irrespective of prior chemotherapy. No more than 3 prior treatment therapies for castration resistant disease (life prolonging) are permitted. Prior therapy can include:

  * Second generation AR targeted therapy (i.e. abiraterone, enzalutamide, or other new antiandrogen [ODM-201, apalutamide])
  * Chemotherapy (docetaxel and/or cabazitaxel)
* Documented progressive mCRPC based on at least one of the following criteria:

  * PSA progression defined as 25% increase over baseline value with an increase in the absolute value of at least 2.0 ng/mL that is confirmed by another PSA level with a minimum of a 1 week interval and a minimum PSA of 2.0 ng/mL
  * Progression of bi-dimensionally measurable soft tissue or nodal metastasis assessed within one month prior to registration by a CT scan or MRI
  * Progression of bone disease (evaluable disease) (new bone lesion[s]) by bone scan
* Serum testosterone < 50 ng/dL. Patients must continue primary androgen deprivation therapy (ADT) with a luteinizing hormone-releasing hormone (LHRH) analogue (agonist or antagonist) if they have not undergone orchiectomy
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients must have adequate organ and bone marrow function as defined below within 28 days of registration:
* Absolute neutrophil count >= 1,000/mcL (within 28 days of registration)
* Hemoglobin >= 9 g/dL* (within 28 days of registration)

  * Transfusion is allowed as long as patients have not received prior transfusion =< 28 days from registration
* Bilirubin =< 1.5 x institutional upper limit of normal (ULN) except for unconjugated hyperbilirubinemia or Gilbert?s syndrome, who can have total bilirubin < 3.0 mg/dL (within 28 days of registration)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN (=< 5 x ULN if liver metastases present) (within 28 days of registration)
* Serum creatinine =< 2.0 X ULN (upper limit of normal) or creatinine clearance >= 30 mL/minute (using Cockcroft/Gault formula) (within 28 days of registration)
* Platelet >= 100,000 (within 28 days of registration)
* Patients must use a condom during treatment and for 3 months after the last dose of study treatment when having sexual intercourse. Female partners of male subjects should also use a highly effective form of contraception if they are of childbearing potential. Subjects should not donate sperm throughout the study and for 3 months following the last dose of treatment
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients who have received more than 3 prior treatment therapies (life prolonging) for mCRPC are not eligible
* Patients who have had radiotherapy =< 14 days prior to entering the study are not eligible

  * Note: Palliative radiation therapy is allowed
* Patients who have had systemic therapy for prostate cancer =< 21 days or 5-half lives (whichever is shorter) are not eligible

  * Note: Patients can receive a stable dose of bisphosphonates for bone metastases, including zoledronic acid, or denosumab before and during the study as deemed appropriate by the treating physician. Patients must continue androgen deprivation therapy
* Patients receiving any other investigational agents are not eligible
* Patients with small cell carcinoma of the prostate are not eligible

  * Note: Neuroendocrine differentiation is permitted. If there is doubt about this and it is clinically indicated then a biopsy should be obtained to document histological differentiation
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to sEphB4-HSA are not eligible. AND patients who have had prior exposure to compounds of similar chemical or biologic composition to sEphB4-HSA are not eligible
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure (New York Heart Association class III or IV congestive heart failure)
  * Unstable angina pectoris
  * Serious cardiac arrhythmia
* Patients with uncontrolled hypertension (defined as systolic blood pressure [BP] >= 160 mmHg or diastolic BP >= 95 mmHg) are not eligible

  * Note: Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
* Patients with electrocardiogram (ECG) with QT interval (corrected QT interval [QTc]) > 480 msec are not eligible
* Patients with other malignancy that has progressed or has required active systemic treatment in the last 3 years

  * Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or carcinoma in situ or non-muscle invasive bladder cancer are not excluded
* Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis are not eligible

  * Note: A scan to confirm the absence of brain metastases is not required. Subjects with previously treated brain metastases may participate provided they are stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), without requirement of steroid treatment for at least 4 weeks prior to randomization and with any neurologic symptoms resolved or have returned to baseline of prior treatment for brain metastasis
* Patients with spinal cord compression are not eligible unless considered to have received definitive treatment for this and evidence of stable disease for 28 days
* Patients who underwent major surgery =< 14 days of starting study treatment or have not recovered from effects of surgery are not eligible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2022-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Maha H Hussain, M.D., Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois

REFERENCES:
- [Derived] VanderWeele DJ, Kocherginsky M, Munir S, Martone B, Sagar V, Morgans A, Stadler WM, Abdulkadir S, Hussain M. A Phase II Study of sEphB4-HSA in Metastatic Castration-Resistant Prostate Cancer. Clin Genitourin Cancer. 2022 Dec;20(6):575-580. doi: 10.1016/j.clgc.2022.08.012. Epub 2022 Sep 7. PMID 36210299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient started treatment on 10/01/2019. The study was designated to enroll patients s with mCRPC who have progressive disease despite castrate levels of testosterone (<50 ng/dL) and have received at least one standard first-line therapy for metastatic castrate resistant prostate cancer, which can include therapy with a 2 nd generation AR targeted therapy (abiraterone or enzalutamide) or chemotherapy (docetaxel or cabazitaxel).The study was closed to further enrollment on 04/07/2021.
Groups:
- Treatment: Patients receive recombinant EphB4-HSA fusion protein IV over 60 minutes on day 1. Treatment repeats every 14 days for cycles 1-6 and then every 21 days for subsequent cycles. Patients may continue to receive sEphB4-HSA treatment until no longer clinically benefiting (PCWG3), unacceptable toxicity, treatment delay >= 4 weeks, or prohibitive illness/change in patient?s condition, or patient decides to withdraw from study.
  Recombinant EphB4-HSA Fusion Protein: Given IV
Period: Overall Study
Arm/Group | Treatment
Started | 14
Registered for Study | 14
Started Cycle 1 | 14
Started Cycle 2 | 13
Started Cycle 3 | 10
Started Cycle 4 | 7
Started Cycle 5 | 1
Started Cycle 6 | 1
Started Cycle 7+ (Beginning at Cycle 7, cycle length will be 21 days and patients will return for treatment on Day 1 of each cycle.) | 1
Completed | 1
Not Completed | 13
Not completed — Progressive Disease | 8
Not completed — Adverse Event | 4
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 14
Age, Customized [Count of Participants; unit: Participants]
  Age: 18-49 | 0
  Age: 50-59 | 2
  Age: 60-69 | 4
  Age: 70-79 | 6
  Age: 80-89 | 2
  Age: 90+ | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Response Rate
Description: Assessment of confirmed PSA response rate is the proportion of subjects who received at least 1 dose of the study drug achieving a post-treatment PSA partial response or complete response as defined by PSA response criteria.
  PSA response criteria:
  These definitions are intended to characterize the PSA changes on study for the purpose of reporting of results.
  Complete Response (CR): Undetectable PSA (<0.2 ng/ml) that is confirmed by another PSA level at no less than 4 weeks interval (+/- 3 days).
  Partial Response (PR): Decrease in PSA value by > 50% that is confirmed by another PSA level at no less than 4 weeks interval (+/- 3 days).
  Stabilization(SD): Patients who do not meet the criteria or PR or PD for at least90 days on the study will be considered stable
  Progression (PD): 25% increase over baseline or nadir whichever is lower and an increase in the absolute value of PSA level by2 ng/ml that is confirmed by another PSA level at no less than 4 weeks interval.
Time Frame: Up to 1 year
Population: From the 14 patients whose PSA data was provided, 14 patients in the sample met the criteria to be assessed for PSA response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Recombinant EphB4-HSA Fusion Protein)
Number analyzed (Participants) | 14
Participants
  Progressive Disease | 13
  Non-Evaluable | 1

2. Secondary Outcome: Incidence of Adverse Events
Description: Will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and reported by the toxicity, severity, and attribution will be recorded for each cycle. All reported adverse event (AE) types will be tabulated by maximum grade using frequencies and percentages. Data on type, timing, frequency and attribution of AEs will also be summarized.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 14
Participants | 14

3. Secondary Outcome: Time to PSA Progression
Description: The time to PSA progression will be assessed by calculating the interval from administration of the first dose of drug on cycle 1 day 1 to PSA progression. PSA progression is defined by the criteria. PSA will be assessed every odd cycle. Will use Kaplan Meier methods to estimate the distribution of time to PSA progression. Will estimate the median with two-sided 90% confidence interval (CI).
Time Frame: From the start of study treatment to PSA progression, assessed for up to 1 year
Population: Of the 14 eligible patients, 14 experienced disease progression by the end of their participation in the study, where progression included events as indicated by PSA values or with a known outcome of death by the time of follow-up. In accordance with the study protocol, a median value for days to progression.
  was calculated along with the 95% confidence interval.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Treatment
Number analyzed (Participants) | 14
Days | 28 [28 to 64]

4. Secondary Outcome: Overall Response Rate
Description: The overall response rate will be the proportion of patients with measurable disease who received at least 1 dose of the study drug and as their best response achieved a partial or complete response (responder). Will be measured according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and PCWG3 criteria. Will be reported with two-sided 90% exact binomial CI.
Time Frame: Up to 1 year
Population: From the 14 patients whose RECIST data was provided, 3 patients in the sample met the criteria to be assessed for RECIST response (receive at least one dose of treatment, have measurable disease). Of the 3 eligible patients, 1 reported tumor progression as his best overall response while 2 patients experienced stabilization as their best overall response. No best overall responses were categorized as partial or complete drug response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 3
Participants
  Stable Disease | 2
  Progressive Disease | 1

5. Secondary Outcome: Time to Radiologic Progression (rPFS)
Description: The time to rPFS will be assessed by calculating the interval from administration of the first dose of drug on cycle 1 day 1 to the time to radiologic progression by RECIST 1.1 or PCWG3 bone criteria or death from any cause. Radiologic assessment will be every 8 weeks. Will use Kaplan Meier methods to estimate the distribution of rPFS. Will estimate the median with two-sided 90% confidence interval (CI).
Time Frame: From the start of study treatment to the time of radiologic progression or death from any cause, assessed for up to 1 year
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Treatment (Recombinant EphB4-HSA Fusion Protein)
Number analyzed (Participants) | 14
Days | 55 [55 to NA] — insufficient number of participants with events

6. Other Pre Specified Outcome: Changes in EphB4 and ephrinB2 Expression
Description: EphB4 and ephrinB2 expression will be assessed by immunohistochemistry (IHC) staining of primary and/or metastatic site (recent archival specimen or new biopsy). EphB4 and other biomarker abnormalities will be assessed by next generation sequencing of metastatic tissue. Will explore if PSA response is associated with expression of EphB4 and ephrinB2 in archival metastatic and primary tumor CRPC specimens. Summaries will be descriptive and graphical.
Time Frame: Baseline up to 1 year
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Circulating Tumor-derived Deoxyribonucleic Acid (ctDNA) Analysis of PI3K Pathway, MYC or TP53
Description: ctDNA will be analyzed for abnormalities in PI3K pathway, MYC or TP53. Summaries will be descriptive and graphical.
Time Frame: Up to 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Immune Infiltrate Characterization in Tumor Specimen
Description: The study will use IHC for CD3, CD4, CD8, and natural-killer cell markers to characterize the immune infiltrate in tumor specimen.
Time Frame: Up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All events that occurred from the day the patient signs consent to within 30 days of the last dose of protocol treatment were reported accordingly. Any event that occurred more than 30 days after the last dose of treatment and is attributed (possibly, probably, or definitely) to the agent(s) must also be was also to be reported accordingly.
Groups:
- Treatment: Patients receive recombinant EphB4-HSA fusion protein IV over 60 minutes on day 1. Treatment repeats every 14 days for cycles 1-6 and then every 21 days for subsequent cycles. Patients may continue to receive sEphB4-HSA treatment until no longer clinically benefiting (PCWG3), unacceptable toxicity, treatment delay >= 4 weeks, or prohibitive illness/change in patient's condition, or the patient decides to withdraw from the study.
  Recombinant EphB4-HSA Fusion Protein: Given IV
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 2/14
Serious Adverse Events (participants affected / at risk) | 3/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=14)
Hematuria (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac troponin I increase (Investigations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=14)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphate increase (Investigations) | 9 (12)
Anaphylaxis (Immune system disorders) | 1 (1)
Anemia (Cardiac disorders) | 7 (11)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood bicarbonate decrease (Investigations) | 2 (2)
Blood bilirubin increase (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fusion Complexes (EKG) (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6)
Creatinine increase (Investigations) | 3 (5)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Dizziness (Nervous system disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Fatigue (General disorders) | 11 (13)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (18)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 13 (36)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (10)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 6 (7)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Anion gap decrease (Investigations) | 1 (1)
Localized edema (General disorders) | 1 (1)
Lymphocyte count decrease (Investigations) | 9 (15)
Malaise (General disorders) | 1 (1)
Mucositis Oral (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Periorbital edema (Eye disorders) | 1 (1)
Platelet count decrease (Investigations) | 5 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Pyuria (Renal and urinary disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus Tachyardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Stroke (Nervous system disorders) | 1 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Weight loss (Infections and infestations) | 4 (6)
White blood cell decrease (Investigations) | 4 (6)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT04033432/Prot_SAP_000.pdf